CLINICAL TRIAL: NCT03070158
Title: Efficacy of a Nursing Intervention in the Mother-premature Infant Affective Bond
Brief Title: Affective Bonding in Mothers and Their Premature Newborn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Industrial de Santander (Other)
Responsible Party: Principal Investigator, Beatriz Villamizar Carvajal, Principal Investigator, Universidad Industrial de Santander
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1900
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Premature Infant
Keywords: Premature Infant; Mother-Infant Interaction; Acoustic stimulation/methods; Touch; Visual Stimulation; Vestibule, Labyrinth/physiology
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The assignment of the mothers to each group will be like that: First at all, mother will be assignment to control group. They will received usual care when achieve the total of 74 mothers, the mothers will be assigned to intervention group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attachment Promotion Intervention (Experimental): Mothers will receive the intervention which includes an education session about newborn care, training in multisensory stimulation with the intervention ATVV and two domiciliary visits to follow up the mother and her premature infant.
  Interventions: Behavioral: Attachment Promotion
- Usual Care (No Intervention): Mothers will continue to receive usual which consist in education session about newborn care in home.

INTERVENTIONS:
Behavioral: Attachment Promotion — Attachment Promotion consists of:
  1. Education session about newborn and mother care.
  2. Training in multisensory stimulation using the ATVV Intervention (auditory, tactile, visual and vestibular)
  3. Two domiciliary visits to follow up and to give education about newborn care and ATVV Intervention.
  4. Daily Phone follows up.
  Arms: Attachment Promotion Intervention

SUMMARY:
This experimental study will determine the effectiveness of nursing intervention "the attachment promotion" to increase the affective bonds between mothers and their premature infants. The assignment of the mothers to the control group will receive usual care, the mothers will be assigned to intervention group will receive the intervention.

DETAILED DESCRIPTION:
The premature newborn has a high need for positive interactions, which is a challenge for him, due to biological immaturity, and for his mother because of the level of stress that this situation generates. Behavioral and developmental interventions are needed to address the unique behaviors of preterm infants and the interactive capacities of the mother-newborn premature dyad. The project will be conducted in 18 months. The assignment of the mothers to each group will be like that: First at all, mother will be assignment to control group. They will received usual care when achieve the total of 74 mothers, the mothers will be assigned to intervention group.

ELIGIBILITY:
Inclusion Criteria:

Premature Infant:

* Neonates who had been hospitalized in the neonatal care unit, with ages ranging from 29 - 36.6/7 weeks gestation at birth.
* Apgar to the minute and five minutes greater to 7/10

Mother:

* Mother with nursing diagnosis: Risk of impaired attachment.
* Mother with a neonate who had hospitalized in the neonatal care unit, with ages ranging from 29 - 36.6/7 weeks of gestation at birth
* Mother living in the metropolitan perimeter of the city of Bucaramanga

Exclusion Criteria:

Newborn:

* Infants that underwent surgery
* Infants with neurological injury.
* Congenital cardiac abnormalities, severe deformities, grade III intraventricular hemorrhage.

Mother:

* Mother with limitations: hearing, motor and / or mental handicap-measured through the Abbreviated Mental Test (minimental), that prevent the intervention.
* Mother consuming psychoactive substances.
* With mental alterations, verified in the medical history.

Ages: 29 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Affective bonding score | 1-6 weeks
  Changes in the mean score of the nursing outcome: affective bonding measure with the NOC(Nursing Outcomes Classification)

SECONDARY OUTCOMES:
Coping adaptation score | 1-6 weeks
  Changes in the mean score of the coping measure with the Coping adaptation Processing Scale Abbreviated (CAPS Abbreviated - Spanish)

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Villamizar- Carvajal, PhD, Principal Investigator — Universidad Industrial de Santander; Carolina Vargas- Porras, Msc, Study Chair — Universidad Industrial de Santander; Mayut Delgado-Galeano, Msc, Study Chair — Universidad Industrial de Santander
Locations (3):
- Colombia (3):
  - Nursing School, Universidad Industrial de Santander, Bucaramanga, Santander Department
  - Clinica Materno Infantil San Luis, Bucaramanga, Santander Department
  - Hospital Universitario de Santander, Bucaramanga, Santander Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Femitha P, Bhat BV. Early neonatal outcome in late preterms. Indian J Pediatr. 2012 Aug;79(8):1019-24. doi: 10.1007/s12098-011-0620-9. Epub 2011 Dec 10. PMID 22161578
- [Background] Kelly MM. Comparison of functional status of 8- to 12-year-old children born prematurely: an integrative review of literature. J Pediatr Nurs. 2012 Aug;27(4):299-309. doi: 10.1016/j.pedn.2011.03.010. Epub 2011 May 11. PMID 22703676
- [Background] Pickler RH, McGrath JM, Reyna BA, McCain N, Lewis M, Cone S, Wetzel P, Best A. A model of neurodevelopmental risk and protection for preterm infants. J Perinat Neonatal Nurs. 2010 Oct-Dec;24(4):356-65. doi: 10.1097/JPN.0b013e3181fb1e70. PMID 21045616
- [Background] Howland LC, Pickler RH, McCain NL, Glaser D, Lewis M. Exploring biobehavioral outcomes in mothers of preterm infants. MCN Am J Matern Child Nurs. 2011 Mar-Apr;36(2):91-7. doi: 10.1097/NMC.0b013e318205587e. PMID 21350371
- [Background] Forcada-Guex M, Borghini A, Pierrehumbert B, Ansermet F, Muller-Nix C. Prematurity, maternal posttraumatic stress and consequences on the mother-infant relationship. Early Hum Dev. 2011 Jan;87(1):21-6. doi: 10.1016/j.earlhumdev.2010.09.006. Epub 2010 Oct 15. PMID 20951514